CLINICAL TRIAL: NCT00078234
Title: A Pilot Study of Genasense® (G3139, Oblimersen Sodium, Bcl-2 Antisense Oligonucleotide), Fludarabine and Rituximab in Previously Treated Subjects With Chronic Lymphocytic Leukemia
Brief Title: Genasense® (Oblimersen Sodium), Fludarabine, and Rituximab in Subjects With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GL217
Record Dates: First submitted 2004-02-20; First posted 2004-02-23 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2009-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; Leukemia; Chronic; Cancer; Adult; Lymphocytic; Genasense; G3139; Genta; Bcl-2; Antisense; Oligonucleotide; oblimersen
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Bronchiolitis Obliterans Syndrome; Neoplasms

INTERVENTIONS:
Drug: Oblimersen-rituximab-fludarabine — 28-day cycles; Cycle 1: oblimersen by continuous IV infusion 1.5 mg/kg/d for 7 consecutive days, completing on Day 8; rituximab by IV infusion on Day 4 (125 mg/m2) and Day 6 (250 mg/m2); fludarabine 25 mg/m2 by IV infusion for 3 days, starting on Day 6. Subsequent cycles: oblimersen 3 mg/kg/d, completing on Day 8; rituximab 375 mg/m2 on Day 5; fludarabine 25 mg/m2 for 3 days starting the same day as rituximab

SUMMARY:
The treatment combination of Rituxan® (rituximab) and fludarabine has previously been reported to produce a high percentage of responses with less toxicity than other combination treatments. However, some leukemia subjects continue to have leukemia despite treatment with these standard anticancer drug therapies, or they may work for only a short period of time. In some subjects, when the leukemia does not respond well to therapy the leukemia cells may be over-producing one or more proteins. One of these proteins is called Bcl-2. Bcl-2 is a protein that appears to protect cancer cells from being killed and thus lengthens the life of the cancer cells. Genasense® (oblimersen sodium) is a compound that blocks production of the Bcl-2 protein. By first lowering levels of Bcl-2, it is possible that chemotherapy drugs may work more effectively as a cancer treatment. Genasense® may also directly kill CLL cells. This study will test whether treating subjects with Genasense®, fludarabine and rituximab is safe and effective.

ELIGIBILITY:
Key Inclusion Criteria:

* Absolute lymphocyte count of > 10,000 cells/mm3 or history of ALC >10,000 cell/mm3
* Platelets > 50,000 cells/mm3
* Tumor lymphocytes expressing surface CD5, CD19, CD20 and CD23
* Creatinine < 1.5 mg.dL

Key Exclusion Criteria:

* Less than 3 weeks from any prior major surgery or other therapy for CLL including radiation therapy, chemotherapy, high-dose steroid therapy, immunotherapy, cytokine, biologic or vaccine therapy.
* History of autoimmune hemolytic anemia
* Prior allogeneic transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-11; Primary Completion 2008-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety and complete response rate | Monthly for response

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Georgetown University Medical Center/Lombardi Cancer Center, Washington D.C., District of Columbia
  - Roswell Park Cancer Institute, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York